CLINICAL TRIAL: NCT05630742
Title: Quality of Life Analysis in Bladder Pain Syndrome/Interstitial Cystitis: Implications for a Multimodal Integrated Treatment
Brief Title: Quality of Life Analysis in Bladder Pain Syndrome/Interstitial Cystitis
Acronym: BPS/IC
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Daniele Porru, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: quality of life in IC
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Interstitial Cystitis, Bladder Pain Syndrome, Quality of Life
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interstitial Cystitis: patients with an existing diagnosis of BPS/IC. BPS/IC was confirmed by reviewing medical record.
- control group: patients with chronic non-neoplastic pain, suffering from fibromyalgia or other types of chronic pain (chronic arthralgia or lower back pain).
  Interventions: Other: chronic non-neoplastic pain

INTERVENTIONS:
Other: chronic non-neoplastic pain — comparison of questionnaires scores
  Groups: control group

SUMMARY:
The aim of our study was to evaluate whether there is a higher prevalence of anxiety-depressive disorders in women with interstitial cystitis than in women with chronic non-neoplastic pain with or without fibromyalgia, to examine possible correlations between urological and psychiatric symptoms, analyze how urological symptoms affect psychological dimension, and how specific stress or trauma can contribute to the onset of interstitial cystitis.

DETAILED DESCRIPTION:
The survey included 69 patients, 42 patients had a diagnosis of Bladder Pain Syndrome/Interstitial Cystitis while 27 of them had chronic non-neoplastic pain. The comparison of the total values of the PHQ-9 between the two groups, 1 versus 2, in relation to final score of PHQ-9, the average PHQ-9 score was 10.3 in group 1, therefore a value greater than 9, considered as major depression (score between 10 and 14); the average score of PHQ-9 was 6.9 in group 2, as in sub-threshold depression (between 5-9). Correlation between PHQ-9 and BPI was also evaluated, the relation was significant only in interstitial cystitis with regard to the following spheres: daily life, work activity, pleasure of life, mood, sleep quality, pain intensity, and urinary symptoms. Based on these data, when PHQ-9 score increases, and depressive symptoms worsen, there is interference with daily life and work activity, pleasure of living, mood, quality of sleep, perception of intensity of pain and urinary symptoms. Patients who had onset of psychiatric symptoms following diagnosis (both interstitial cystitis and other painful syndromes) had an average PHQ-9 score of 11.7 compared to the score of 8.3 of patients without onset of psychiatric symptoms after diagnosis (p = 0.0464), so it may be that depressive symptoms starting after the diagnosis of pain syndrome are more severe. Women who undergo psychiatric-psychological consultation and therapy have an average O'Leary score 20.4 compared to 25.8 in those who are not under psychiatric consultation (p = 0.0418). This emphasizes how psychosocial support can improve perception of pain and urinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients aged > 18 years diagnosis of BPS/IC or chronic non-neoplastic pain
* Exclusion Criteria:

bladder cancer

-

Ages: 18 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: patients with an existing diagnosis of BPS/IC. We confirmed presence of BPS/IC by reviewing medical record.
  Group 2: patients with chronic non-neoplastic pain, suffering from fibromyalgia or other types of chronic pain (chronic arthralgia or lower back pain).
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
psychological symptoms and perception of pain affect every aspect of patients' life in IC | 9 months
  PHQ-9: to investigate psychological symptoms, O'Leary Saint (ICSI-ICPI) to investigate urological symptoms only for women with I.C and BPI questionnaires were administered
Examine whether there is a higher prevalence of anxiety-depressive disorders in women with interstitial cystitis than in women with chronic non-neoplastic pain with or without fibromyalgia. | 9 months
  PHQ-9: to investigate psychological symptoms, O'Leary Saint (ICSI-ICPI) to investigate

SECONDARY OUTCOMES:
correlations between urological symptoms and psychiatric symptoms | 9 months
  PHQ-9: to investigate psychological symptoms, O'Leary Saint (ICSI-ICPI) to investigate

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Dept. Policlinico an Matteo, Pavia, Pv, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKernan LC, Bonnet KR, Finn MTM, Williams DA, Bruehl S, Reynolds WS, Clauw D, Dmochowski RR, Schlundt DG, Crofford LJ. Qualitative Analysis of Treatment Needs in Interstitial Cystitis/Bladder Pain Syndrome: Implications for Intervention. Can J Pain. 2020;4(1):181-198. doi: 10.1080/24740527.2020.1785854. Epub 2020 Sep 1. PMID 33367196
- [Background] Naliboff BD, Stephens AJ, Afari N, Lai H, Krieger JN, Hong B, Lutgendorf S, Strachan E, Williams D; MAPP Research Network. Widespread Psychosocial Difficulties in Men and Women With Urologic Chronic Pelvic Pain Syndromes: Case-control Findings From the Multidisciplinary Approach to the Study of Chronic Pelvic Pain Research Network. Urology. 2015 Jun;85(6):1319-27. doi: 10.1016/j.urology.2015.02.047. PMID 26099876
- [Result] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797